CLINICAL TRIAL: NCT03272997
Title: The Diagnostic Power of 18F-FDG PET-CT Scanning for Discriminating Malignant From Non-malignant Causes in Unilateral Pleural Effusions
Brief Title: The Value of PET-CT in Pleural Effusions
Status: Completed | Type: Observational
Sponsor: Naestved Hospital (Other)
Responsible Party: Principal Investigator, Simon Reuter, MD, Principal investigator, Naestved Hospital
Other Study IDs: PET-CT in UPE
Record Dates: First submitted 2017-08-30; First posted 2017-09-06 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Pleural Effusion, Malignant
Keywords: Positron emission thomography; Computed tomography; Sensitivity; Specificity
MeSH Terms: conditions — Pleural Effusion, Malignant; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aim is to asses the diagnostic power of 18F-FDG PET-CT in discriminating malignant from nonmalignant causes in patients with a recurrent unilateral pleural effusion of unknown origin.

DETAILED DESCRIPTION:
The investigators follow the STARD 2015 guideline for reporting diagnostic accuracy studies.

The investigators will review the hospital's administrative database of patients who underwent a thoracocentesis from January 2013 to January 2015. Patients at Department of Respiratory Medicine, Zealand University Hospital, Roskilde and Department of Respiratory Medicine, Naestved Hospital, Region Zealand, Denmark (two large respiratory centres with specialised functions) is eligible for inclusion. Patients are included irrespective of cytology and chemical analysis.

The investigators will review the patients' medical records and images retrospectively. To reduce the number of false negatives, the investigators complete a 1-year follow-up.

Patients older than 16 years are included, irrespective of smoking history and comorbidities, if both thoracocenteses, chest x-ray, a CT-scanning and a PET-CT scanning is performed. Exclusion criteria are previously diagnosed lung cancer, thoracic malignancy or incomplete data.

Classification of results The investigators chose the combination of investigations recommended by the internationally acknowledged BTS guideline, which is endorsed by the Danish Society of Respiratory Medicine. Thoracocentesis, chest x-ray, CT findings and PET-CT findings is categorized as either normal (i.e. not suggestive of any aetiology of the unilateral pleural effusion), suggestive of other lung pathology or suggestive of malignancy (i.e. representing a possible aetiology of the unilateral pleural effusion).

The thoracocentesis is classified as malignant if cytological examination revealed malignant cells. The chest x-ray is classified as malignant if suspicion of malignant disease is not rejected. The CT findings are classified as malignant according to Leung et. al. for pleural abnormalities (circumferential pleural thickening, nodular pleural thickening, parietal pleural thickening > 1 cm and mediastinal pleural involvement) and The Fleischner Society for parenchymal abnormalities (nodules > 8 mm). The PET-CT findings are classified as malignant if any findings suspicious for malignancy.

CT and PET-CT images, as well as the scan reports by the radiologist and the nuclear medicine physician, is reviewed by two experienced pulmonologists. They are blinded to all patient information, including final diagnosis.

The final diagnosis, the reference standard, is extracted from the patients' medical records. When no diagnosis is found, two investigators agree on a consensus diagnosis based on all investigation results. If no reasonable diagnosis can be established based on the findings, the patient case is categorized as having no final diagnosis. These cases are treated as a worst-case scenario, i.e. patients with a malignant disease are treated as false negative, and patients without malignant disease are treated as false positive.

Statistics Data are presented as frequencies and/or mean ± standard deviation (SD). Test characteristics were compared using McNemar's test with Bonferroni correction (two-sided level of significance < o.o5). Diagnostic power of thoracocentesis, chest x-ray, CT-scanning, PET-CT scanning and the combination are calculated. Diagnostic power is defined as true positive, true negative, false positive, false negative, sensitivity, specificity, likelihood ratio+, likelihood ratio-, positive predictive value (PPV), negative predictive value (NPV) and diagnostic accuracy (TP+TN)/(TP+FP+TN+FN).

The combined sensitivity will be calculated using the formula:

Sensitivitytest A + Sensitivitytest B + Sensitivitytest … - (Sensitivitytest A x Sensitivitytest B x Sensitivitytest …)

The combined specificity will be calculated using the formula:

Specificitytest A x Specificitytest B x Specificitytest… Data were analyzed using STATA (StataCorp LLC, Version 15.0, College Station, Texas, USA).

ELIGIBILITY:
Inclusion Criteria:

* Thoracocentesis
* Chest X-ray
* CT scanning
* PET-CT scanning

Exclusion Criteria:

* Missing data
* Lung cancer
* Thoracic malignancies

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a unilateral pleural effusion of unknown origin examined with the above
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity PET-CT | 1 year
  TP / (TP + FN)

SECONDARY OUTCOMES:
CT-Specificity | 1 year
  TN / (TN+FP)
PET-CT-Specificity | 1 year
  TN / (TN+FP)
CT-Sensitivity | 1 year
  TP / (TP + FN)
Comparison of the diagnostic power | 1 year
  McNemars' test with Bonferroni
CT-Likelihood ratio+ | 1 Year
  LR+ = sensitivity / (1-specificity)
PET-CT-Likelihood ratio+ | 1 Year
  LR+ = sensitivity / (1-specificity)
CT-Likelihood ratio- | 1 year
  LR- = (1-sensitivity) / specificity
PET-CT-Likelihood ratio- | 1 year
  LR- = (1-sensitivity) / specificity
CT-positive predictive value | 1 year
  PPV =TP / (TP+ FP)
PET-CT-positive predictive value | 1 year
  PPV =TP / (TP+ FP)
CT-negative predictive value | 1 year
  TN/ (TN + FN)
PET-CT-negative predictive value | 1 year
  TN/ (TN + FN)
CT-Diagnostic accuracy | 1 year
  (TP+TN) / (TP+TN+FP+FN)
PET-CT-Diagnostic accuracy | 1 year
  (TP+TN) / (TP+TN+FP+FN)

CONTACTS AND LOCATIONS:
Locations (1):
- Naestved Hospital, Næstved, Denmark